CLINICAL TRIAL: NCT03446404
Title: Standing Computerized Tomography (SCT) Imaging of the Knee Joint in People With or at Risk for Knee Osteoarthritis (KOA)
Brief Title: Standing Computed Tomography (SCT) Imaging of the Knee Joint
Status: Completed | Type: Observational
Sponsor: Neil A Segal (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Sponsor-Investigator, Neil A Segal, Adjunct Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201602741
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- MOST Cohort: One portion of the cohort will be age 62-92 years, average age approximately 71 years, at the start of this study. This cohort will consist of participants who already have symptomatic knee OA, in many cases advanced disease, or who had risk factors at the start of the Multicenter Osteoarthritis Study but have not developed symptomatic knee OA. All of the existing cohort who have 1 or 2 "native" knees will be approached providing native knees are not considered to be Kellgren-Lawrence grade 4 (bone on bone). The other portion of the cohort will consist of subjects with knee pain, aching or stiffness at baseline and participants without any knee symptoms in the previous 30 days. Both knees with Kellgren-Lawrence grades of radiographic OA of 0, 1, or 2 in the tibiofemoral (TF) and patellofemoral (PF) compartments.
  Interventions: Diagnostic Test: Standing Computed Tomography

INTERVENTIONS:
Diagnostic Test: Standing Computed Tomography — Provides weight bearing 3D view of knees.
  Other Names: SCT

SUMMARY:
This study will help us decide the best way to image the knee for diagnostic purposes: Knee computed tomography vs knee x-ray. The computed tomography will provide a weight bearing 3D view.

DETAILED DESCRIPTION:
This will be an ancillary study to the Multicenter Osteoarthritis Study (MOST) second renewal #201511711). Using a prototype Curve Beam Standing Computed Tomography (SCT) scanner to get a 3 dimensional picture of the knee joint, bilaterally. This scanner by Curve Beam 175 Titus Ave, Suite 300, Warrington, Pennsylvania 18976, has been approved by the Food and Drug Administration (FDA) for ankles and feet. This has been modified to do the scan of the knee but is not yet approved by the FDA for the knees. The proposed ancillary study would add the key benefit of providing more sensitive and accurate identification of prevalent knee osteoarthritis (OA) at baseline and incident knee OA at follow-up than is available with plain radiographs. In addition, it would enable biomechanical modeling of the knee joint on a larger scale than achieved in any prior study, allowing testing of biomechanical hypotheses regarding mechanisms of disease development and progression that have not been possible on this scale previously.

ELIGIBILITY:
Inclusion Criteria:

Only participants in the Multicenter Osteoarthritis Study (MOST) who attend a 0/144-month visit at the Iowa site are eligible for inclusion.

Additional Inclusion Criteria Include:

* Completed knee radiograph (posteroanterior view) at 0/144-month visit of primary MOST-second renewal study at the Iowa Site

Exclusion Criteria:

* Bilateral Total Knee Arthroplasty

Ages: 45 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The existing cohort will be age 62-92 years, average age approximately 71 years, at the start of this study. This cohort will consist of participants who already have symptomatic knee OA, in many cases advanced disease, or who had risk factors at the start of MOST but have not developed symptomatic knee OA. All of the existing cohort who have 1 or 2 "native" knees will be approached providing native knees are not considered to be KL grade 4 (bone on bone). The new cohort will consist of subjects with knee pain, aching or stiffness at baseline and participants without any knee symptoms in the previous 30 days. Both knees with KL grades of radiographic OA of 0, 1, or 2 in the tibiofemoral (TF) and patellofemoral (PF) compartments.
Sampling Method: Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Change in Joint Space Width | Baseline and 2-years
  3D measurement of distance between articular surfaces of tibia and femur

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, MS, Principal Investigator — University of Iowa and University of Kansas
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
As an ancillary study to the Multicenter Osteoarthritis Study (MOST), data will be available to other researchers through the MOST Data Sharing Plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following study completion (anticipated August 2021)

REFERENCES:
- [Background] Segal NA, Frick E, Duryea J, Roemer F, Guermazi A, Nevitt MC, Torner JC, Felson DT, Anderson DD. Correlations of Medial Joint Space Width on Fixed-Flexed Standing Computed Tomography and Radiographs With Cartilage and Meniscal Morphology on Magnetic Resonance Imaging. Arthritis Care Res (Hoboken). 2016 Oct;68(10):1410-6. doi: 10.1002/acr.22888. PMID 26991547
- [Background] Segal NA, Nevitt MC, Lynch JA, Niu J, Torner JC, Guermazi A. Diagnostic performance of 3D standing CT imaging for detection of knee osteoarthritis features. Phys Sportsmed. 2015 Jul;43(3):213-20. doi: 10.1080/00913847.2015.1074854. Epub 2015 Aug 3. PMID 26313455
- [Background] Segal NA, Stockman TJ, Findlay CM, Kern AM, Ohashi K, Anderson DD. Effect of a Realigning Brace on Tibiofemoral Contact Stress. Arthritis Care Res (Hoboken). 2015 Aug;67(8):1112-8. doi: 10.1002/acr.22578. PMID 25779857
- [Background] Sheehy L, Culham E, McLean L, Niu J, Lynch J, Segal NA, Singh JA, Nevitt M, Cooke TD. Validity and sensitivity to change of three scales for the radiographic assessment of knee osteoarthritis using images from the Multicenter Osteoarthritis Study (MOST). Osteoarthritis Cartilage. 2015 Sep;23(9):1491-8. doi: 10.1016/j.joca.2015.05.003. Epub 2015 May 21. PMID 26003948
- [Background] Stefanik JJ, Gross KD, Guermazi A, Felson DT, Roemer FW, Zhang Y, Niu J, Segal NA, Lewis CE, Nevitt M, Neogi T. The relation of MRI-detected structural damage in the medial and lateral patellofemoral joint to knee pain: the Multicenter and Framingham Osteoarthritis Studies. Osteoarthritis Cartilage. 2015 Apr;23(4):565-70. doi: 10.1016/j.joca.2014.12.023. Epub 2015 Jan 7. PMID 25575967